CLINICAL TRIAL: NCT04248062
Title: Identification and Validation of Relevant Patient and Observer Reported Outcome Measurements in Inborn Errors of Metabolism
Brief Title: Patient and Observer Reported Outcome Measurements in Inborn Errors of Metabolism
Acronym: MetaPROM
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 10650
Record Dates: First submitted 2019-11-07; First posted 2020-01-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Inborn Errors of Metabolism; Urea Cycle Disorder; Maple Syrup Urine Disease; Phenylketonurias; Methylmalonicacidemia; OTC Deficiency; Aminoacidopathy; Patient Reported Outcome Measurements
MeSH Terms: conditions — Metabolism, Inborn Errors; Urea Cycle Disorders, Inborn; Maple Syrup Urine Disease; Phenylketonurias; Methylmalonic acidemia; Ornithine Carbamoyltransferase Deficiency Disease; Amino Acid Metabolism, Inborn Errors | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IEM experts: Heterogeneous group of health professionals (physicians, psychologists, nutritionists) working in the field of Inborn Errors of Metabolism (IEM)
  Interventions: Other: Survey
- Paediatric IEM patients: IEM patients between 10 and 18 years
  Interventions: Other: Survey
- Parents of paediatric IEM patients and patient representatives: * Parents of IEM patients (between 0 and 18 years)
  * Patient representatives
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey: 38 preselected patient and parent reported outcomes; rating scale: 9 point likert scale (1=not at all important - 9=very important)

SUMMARY:
lnborn errors of metabolism (IEM) are a heterogeneous group of rare, sometimes debilitating or even fatal diseases . In IEM, both definition and assessment of meaningful outcome parameters is often extremely difficult resulting in a limited body of evidence. Limited evidence results in weak recommendations which are perceived as unbinding and thus sustains heterogeneous study designs, choice of outcomes and interventions again producing non-uniform data.

The goal of the current study is to identify and select reliable instruments, that measure patients' and their parents' perception about relevant (social, emotional, cognitive and physical) aspects in their lives. This set of instruments will secure the comparability of future research findings. Furthermore this instruments will improve the screening of paediatric IEM patients regarding their need for additional (psychosocial or consultative) support in daily hospital routine.

DETAILED DESCRIPTION:
1. Background

   Limitations to the body of evidence on effects of interventions on important outcome parameters in IEM and thus to evidence-based recommendations or guidelines are manifold. Due to the rarity of each disease, knowledge about the natural history may be poor. Most IEM are clinically heterogeneous with severity of the disease determined by mutation type, residual enzyme activity and additional, often unidentified factors. Consecutively, studies in IEM are variable regarding outcome parameters, treatment regimens and targets. Often the evidence on meaningful outcomes is scarce because only small subgroups of studies address them in a structured and standardized manner. In IEM, there is a long-standing preference for biochemical outcome parameters, such as for example phenylalanine (Phe) concentrations in phenylketonuria or total homocysteine levels in patients with remethylation disorders. However, even these at first glance objective outcome parameters have their drawbacks: Phe targets differ significantly between countries and for the remethylation disorders there is no general agreement on precise target ranges for total homocysteine. Due to these circumstances, studies set different targets. Moreover, for same IEM no meaningful biochemical parameters are even available (e.g. Pompe disease). More and more Patient-reported outcome measures are recognized as valid additional, complementary parameters for evaluating pharmacological, dietary or disease-management interventions in chronic diseases. PROMs are directly reported by the patient (and their parents). PROMs can be used as single measurements to assess the patient's current situation or to report changes from a previous measure (e.g. following an Intervention). In contrast to the well-established parameters such as biochemical markers or disease-related mortality, PROMs allow direct insight into experience and performance of a patient and / or his caregivers in everyday life. Furthermore, use of PROMs in the clinical setting improves survival rates as well as patients' satisfaction with care, disease management as well as health-related quality of life (HrQoL).
2. Current study

In the current study the relevance of patient reported outcomes (PROs) for paediatric IEM patients and their families will be identified via Delphi method. 35 IEM experts (physicians, psychologists, nutritionists) and 30 patients and parents (anticipated 15 patients / 15 parents) will fill out a survey including potentially relevant aspects of life in paediatric IEM (preselected by the interdisciplinary research team based on conducted focus groups in a previous study). Participants will be asked to rate every PRO regarding their relevance. A second survey, including only the important aspects (criteria based on Delphi manuals), will then be completed by the participants, to reach further deduction. Afterwards, a focus group with participants of the two surveys (6 metabolic experts / 3 parents / 3 patients > 12 years) will be held at the University Children's Hospital in Zurich, to discuss unclear ratings and additional PRO suggestions. For the remaining PROs, corresponding PROMs will be selected by the interdisciplinary research team based on the criteria of reliability, (face-, construct-) validity, quality of norm data, and frequency of usage in research.

ELIGIBILITY:
*Statements above refer to IEM patients included in the study

Inclusion Criteria (patients):

* Suffering from rare IEM (e.g. phenylketonuria, urea cycle disorders, maple syrup urine disease, methylmalonic acidemia)
* Ability to understand German language
* Cognitive ability to complete the basic survey items

Inclusion Criteria (parents):

* Ability to understand German language
* Parents of a child suffering from IEM

Inclusion Criteria (experts):

* More than 1 year of practical experience in the field of IEM
* Ability to understand written English

Exclusion Criteria (patients):

* Older than 18 years
* Severe cognitive impairment (ability to complete the Survey not existent)

Inclusion Criteria (parents):

* No ability to understand German language

Exclusion Criteria (experts):

* Less than 1 year of practical experience in the field of IEM
* No ability to understand written English

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The included groups (experts, patients, parents/patient representatives) were all not randomly chosen.
  Experts are recruited based on the criteria of profession, specialization, experience and location. A sample as balanced as possible is intended.
  Patients and their parents are recruited based on IEM disease, disease severity, age and gender. A sample as balanced as possible is intended.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Average importance of patient reported outcomes (PRO) after first Delphi survey | 15 minutes (for Delphi survey 1)
  Average importance-rating of the PROs in the total sample (experts, patients, parents, patient representatives); 9-point Likert scale (1 = not at all important, 2 = very important); Sum-Score for each PRO divided by number of survey-participants; Consensus about the importance of a PRO achieved if at least 70% of the voting participants from each stakeholder group scored between 7 and 9
Average importance of patient reported outcomes (PRO) after second Delphi survey | 15 minutes (for Delphi survey 2)
  Average importance-rating of the PROs in the total sample (experts, patients, parents, patient representatives); 9-point Likert scale (1 = not at all important, 2 = very important); Sum-Score for each PRO divided by number of survey-participants; Consensus about the importance of a PRO achieved if at least 70% of the voting participants from each stakeholder group scored between 7 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Martina Huemer, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
In the scheduled publication, sharing of individual's voting data is not planned. The investigator's research interest refers to the average importance-voting regarding the preselected PROs.

REFERENCES:
- [Background] Slade A, Isa F, Kyte D, Pankhurst T, Kerecuk L, Ferguson J, Lipkin G, Calvert M. Patient reported outcome measures in rare diseases: a narrative review. Orphanet J Rare Dis. 2018 Apr 23;13(1):61. doi: 10.1186/s13023-018-0810-x. PMID 29688860
- [Background] Morel T, Cano SJ. Measuring what matters to rare disease patients - reflections on the work by the IRDiRC taskforce on patient-centered outcome measures. Orphanet J Rare Dis. 2017 Nov 2;12(1):171. doi: 10.1186/s13023-017-0718-x. PMID 29096663
- [Background] Zeltner NA, Landolt MA, Baumgartner MR, Lageder S, Quitmann J, Sommer R, Karall D, Muhlhausen C, Schlune A, Scholl-Burgi S, Huemer M. Living with Intoxication-Type Inborn Errors of Metabolism: A Qualitative Analysis of Interviews with Paediatric Patients and Their Parents. JIMD Rep. 2017;31:1-9. doi: 10.1007/8904_2016_545. Epub 2016 Aug 13. PMID 26983835
- [Background] Weldring T, Smith SM. Patient-Reported Outcomes (PROs) and Patient-Reported Outcome Measures (PROMs). Health Serv Insights. 2013 Aug 4;6:61-8. doi: 10.4137/HSI.S11093. eCollection 2013. PMID 25114561